CLINICAL TRIAL: NCT03253120
Title: Alterations of Attention in Patients With Postural Tachycardia Syndrome and Healthy Controls Depending on Body Position and Hydration
Brief Title: Alterations of Attention in POTS Depending on Body Position and Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01368
Record Dates: First submitted 2017-08-02; First posted 2017-08-17 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Postural Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Water

STUDY DESIGN:
Intervention Model Description: Patients will drink 5dl of water. Healthy volunteers will drink 5dl of water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient (Other): Patients will drink 5dl of water.
  Interventions: Other: Water
- Healthy volunteer (Other): Healthy volunteers will drink 5dl of water.
  Interventions: Other: Water

INTERVENTIONS:
Other: Water — Patient/ Healthy volunteer will drink 5dl of Water

SUMMARY:
The Postural Tachycardia-Syndrome (POTS) is a form of autonomic dysregulation, typically accompanied by symptoms of orthostatic intolerance (OI). OI is defined by the inability to tolerate the upright position and is improved by lying down. POTS is considered a syndrome that may include a number of several disorders. Symptoms should be persistent for at least 6 months to reach a diagnosis. It is characterized by a sustained heart rate (HR) increment of 30 beats/min or more within 10 min of standing or head-up tilt (HUT) in adults, in the absence of orthostatic hypotension and with the presence of symptoms of OI. In children and adolescents a diagnosis requests a HR increment of at least 40 beats/min. The increment in HR when moving to an upright posture is often a response to a reduction in venous return, causing excessive blood pooling in the lower limbs. The symptoms present in POTS vary greatly. Typical symptoms are lightheadedness, dizziness, blurred vision, mental clouding ("brain fog") or cognitive dysfunction. Other symptoms may present as palpitations or chest pain. Additional symptoms consist of postural headaches, nausea, sleep disturbances, fatigue and gastrointestinal dysfunction. The manifestation of symptoms in POTS varies in severity, frequency and combination, resulting in POTS being a very heterogenous and subjective disorder. Symptoms can be severe and often make simple daily activities difficult to an extent that compromises the patients quality of life. Typically symptoms exacerbate in the mornings, after physical activity, after eating and during menstruation.

This study objective is to examine the occurrence, mechanisms and causes of impaired attention in POTS as well as to test the effect of acute water ingestion for attention in POTS. The investigators therefore conduct a study including patients with POTS and healthy volunteers.

All participants will receive a dossier of five self-assessment questionnaires after giving informed consent. Clinical examination includes 2 HUT-tests while standing for 15 minutes, conventional measuring of blood pressure, continuous recording of NIRS signals during testing, determination of pupil size, the diameter of the optic nerve and Neuropsychological testing (Test of Attentional Performance, mobility version" (TAP-M), Go/NoGo Test, Divided Attention Test)

DETAILED DESCRIPTION:
Background

Postural Tachycardia Syndrome (POTS) is a form of autonomic dysregulation, typically accompanied by symptoms of orthostatic intolerance (OI). OI is defined by the inability to tolerate the upright position and is improved by lying down. POTS is considered a syndrome that may include a number of several disorders. Symptoms should be persistent for at least 6 months to reach a diagnosis. It is characterized by a sustained heart rate (HR) increment of 30 beats/min or more within 10 min of standing or head-up tilt (HUT) in adults, in the absence of orthostatic hypotension and with the presence of symptoms of OI. In children and adolescents diagnosis requests a HR increment of at least 40 beats/min. The increment in HR when moving to an upright posture is often caused by a reduction in venous return because of excessive blood pooling in the lower limbs. Clinical symptoms present in POTS vary greatly. Typical symptoms are palpitations, lightheadedness, dizziness, blurred vision, mental clouding ("brain fog") or cognitive dysfunction . Additional symptoms consist of postural headaches, nausea, but also non-orthostatic symptoms such as sleep disturbances, fatigue and gastrointestinal dysfunction. The manifestation of symptoms in POTS varies in severity, frequency and combination, resulting in POTS being a very heterogenous and subjective disorder. Symptoms can be severe and make simple daily activities difficult. Typically symptoms exacerbate in the mornings, after physical activity, after eating and during menstruation. The onset of the syndrome is associated with a variety of possible causes, e.g. a recent viral illness or autonomic neuropathy.

As mentioned above, some of the most frequent reported symptoms are concentration- and attentional problems so called "brain fog" or "mental clouding". Previous research indicates an actual deficit in cognitive functioning, which is, same as other POTS symptoms, exclusive to the upright position. However, there is no overall accepted and recognized definition of what "brain fog" is or what components it consists of. The majority of studies examined, amongst other things, aspects of attention and working memory. Ross et al. compared it to mental fatigue and showed that 67% of all POTS patients experience this symptom on a daily basis, which indicates that routine daily activities and consequent quality of life are reduced even further.

Conservative therapy in POTS consists in a high intake of water (2-3L) and salt on a daily basis, wearing compression stockings and regular endurance training. Severely affected patients may profit from additional drug treatment. A previous research group of the investigators' unit showed in 2010 the improvement of OI in POTS after acute water and clear soup intake.

Objective:

The purpose of this study is to examine the occurrence, mechanisms and causes of impaired attention in POTS as well as to test the effect of acute water ingestion for attention in POTS.

The study consists of four different assessments

Methode:

All participants will receive a dossier of five self-assessment questionnaires after giving informed consent. The dossier consists of: Beck's Depression Inventory II (BDI-II) for assessing depression, Short Form (36) Health Survey (SF-36) for assessing health-related quality of life, Pittsburgh Sleep Quality Index (PSQI) for assessing sleep quality, International Physical Activity Questionnaire (IPAQ) for assessing personal physical activity and a questionnaire designed to measure specific symptoms in POTS (POTS Questionnaire) to assess and objectify the symptomatology of POTS patients. The completion is expected to take approximately one hour.

The study consists of four different assessments. For the examination all POTS medication will be stopped prior to the examination. All participants have no dietary restrictions during the days before the study, but will have to ingest nil by mouth after midnight.

For autonomic function testing, beat-to-beat BP and HR are measured (with the Finometer device). At the beginning of each assessment, intermittent brachial BP and HR values will be simultaneously recorded (using an automated Dinamap Pro 100 sphygmomanometer) on the right arm. In addition, continuous recording of NIRS signals during testing will be acquired.

The study will start with a supine rest on an electrical tilt table for at least 10 minutes, whilst BP and HR settle and sufficient correlation between Finometer and Dinamap readings are achieved. A baseline assessment of attention in supine position follows, before tilting the participants to a 60°upright position. In the upright position participants will again perform the same assessment of attention. Patients will be at a tilt angle of 60° for a maximum of 20 minutes. HUT will be terminated earlier in case of pre-syncope. After a short recovery in the supine position, participants will be asked to drink 5 dl of commercially available still mineral water within 5 minutes. To facilitate rapid drinking, the upper body will be transiently elevated for 45-60°. After drinking, participants will again be supine for 20 minutes before a second assessment of attention in the supine position. Subsequently participants will again be tilted to 60° and complete the second assessment of attention in the upright posture. HUT will be terminated earlier in case of pre-syncope. The duration of tolerated HUT at baseline and after fluid ingestion will be noted.

Patients will be asked to rate their experienced symptoms in the upright position both before and after the intake of water.

Neuropsychological testing will consist of three subtests of the automated computer-based test battery "Test of Attentional Performance, mobility version" (TAP-M). Second the investigators will use the "Go/NoGo" task for assessing the specific ability of subjects to suppress undesired responses. Reaction times and errors are recorded in a simple test with two stimuli. Using the subtest of "Divided Attention", deficits of divided attention will be measured, which are frequently diagnosed in neuropsychological practice. This can be assessed in a "dual-task" paradigm, in which two stimuli have to be attended to simultaneously. The test battery is computer-based; the screen will be placed in a distance of 30 cm from the participants face and the button for reaction responses will be held in the dominant hand. For capturing a possible decrease in attentional performance participants will complete the sequence of the three subtests two times in two respective blocks, resulting in a total duration time of 15 minutes.

The diameter of the optic nerve is measured with a 7-15 MHz linear array transducer in transorbital B-mode ultrasound.

The investigators expect a study duration of approximately four hours.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Informed consent
* Patients with diagnosed POTS (for criteria, see above)
* Age: ≥18 years and ≤ 60 years

For healthy volunteers:

* Informed consent
* Age: ≥18 years and ≤ 60 years

Exclusion Criteria:

For patients:

* Pregnancy and Breastfeeding
* Due to clinical reasons the current medication for POTS can not be discontinued

For healthy volunteers:

* Pregnancy and Breastfeeding
* Intake of vasoactive medication or known, non-treated arterial hypertension
* Known vasovagal syncope in medical history

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Numerical variables reaction time and/or hits resp. misses in the subtests "alertness" from the automated test battery "Test of Attentional Performance, mobility version" | After change body position and 5dl of water, up to 30 minutes
  "Alertness" is designed to assess tonic alertness, which is defined as the ability to maintain a high level of responsiveness in anticipation of a test stimulus. The alertness test measures the simple reaction time in response to a visual stimulus (a cross presented on the monitor)
Numerical variables reaction time and/or hits resp. misses in the subtest "Go/NoGo" from the automated test battery "Test of Attentional Performance, mobility version" | After change body position and 5dl of water, up to 30 minutes
  The "Go/NoGo" task for assessing the specific ability of subjects to suppress undesired responses. Reaction times and errors are recorded in a simple test with two stimuli
Numerical variables reaction time and/or hits resp. misses in the subtest "divided attention" from the automated test battery "Test of Attentional Performance, mobility version" | After change body position and 5dl of water, up to 30 minutes
  In the Test of Attentional Performance a visual and an auditory task must be processed in parallel

SECONDARY OUTCOMES:
Diameter of the optic nerve | After change body position and 5dl of water, up to 30 minutes
  The diameter of the optic nerve is measured with a 7-15 MHz linear array transducer in transorbital B-mode ultrasound .
Brain perfusion measured with NIRS | After change body position and 5dl of water, up to 30 minutes
  All parameters of brain perfusion will be assessed using NIRS.
Heart rate | After change body position and 5dl of water, up to 30 minutes
  For autonomic function testing, beat-to-beat BP and HR are measured with the Finometer device.
Blood pressure | After change body position and 5dl of water, up to 30 minutes
  For autonomic function testing, beat-to-beat BP and HR are measured with the Finometer device.
Pupil diameter | After change body position and 5dl of water, up to 30 minutes
  Determination of pupil size will be performed with a rubber cup covering the measured eye and the operator's hand covering the nonmeasured eye. A brief 2- to 3-second pause allows the pupil to dilate briefly at which time the measurement will be taken. Pupil size is the average diameter for the entire measurement time, which is typically 3 to 4 seconds.

OTHER OUTCOMES:
Scores of the questionnaires (composite endpoint) | Through study completion an average of 1 day
  Beck's Depression Inventory II (BDI-II) for assessing depression, Short Form (36) Health Survey (SF-36) for assessing health-related quality of life, Pittsburgh Sleep Quality Index (PSQI) for assessing sleep quality, International Physical Activity Questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Werner Z'Graggen, MD, Principal Investigator — Inselspital Bern, Department of Neurosurgery and Neurology
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson JW, Lambert EA, Sari CI, Dawood T, Esler MD, Vaddadi G, Lambert GW. Cognitive function, health-related quality of life, and symptoms of depression and anxiety sensitivity are impaired in patients with the postural orthostatic tachycardia syndrome (POTS). Front Physiol. 2014 Jun 25;5:230. doi: 10.3389/fphys.2014.00230. eCollection 2014. PMID 25009504
- [Background] Arnold AC, Haman K, Garland EM, Raj V, Dupont WD, Biaggioni I, Robertson D, Raj SR. Cognitive dysfunction in postural tachycardia syndrome. Clin Sci (Lond). 2015 Jan;128(1):39-45. doi: 10.1042/CS20140251. PMID 25001527
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Lambert E, Lambert GW. Sympathetic dysfunction in vasovagal syncope and the postural orthostatic tachycardia syndrome. Front Physiol. 2014 Jul 28;5:280. doi: 10.3389/fphys.2014.00280. eCollection 2014. PMID 25120493
- [Background] Ocon AJ, Messer ZR, Medow MS, Stewart JM. Increasing orthostatic stress impairs neurocognitive functioning in chronic fatigue syndrome with postural tachycardia syndrome. Clin Sci (Lond). 2012 Mar;122(5):227-38. doi: 10.1042/CS20110241. PMID 21919887
- [Background] Raj SR. Postural tachycardia syndrome (POTS). Circulation. 2013 Jun 11;127(23):2336-42. doi: 10.1161/CIRCULATIONAHA.112.144501. No abstract available. PMID 23753844
- [Background] Z'Graggen WJ, Hess CW, Humm AM. Acute fluid ingestion in the treatment of orthostatic intolerance - important implications for daily practice. Eur J Neurol. 2010 Nov;17(11):1370-6. doi: 10.1111/j.1468-1331.2010.03030.x. PMID 20412295